CLINICAL TRIAL: NCT00910975
Title: Tailored Treatment of Hepatitis C Genotype 1
Brief Title: Individualized Duration of Peg-interferon/Ribavirin Treatment of Hepatitis C
Acronym: TTG1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Sodra Alvsborgs Hospital (Other); Skaraborg Hospital (Other Government); Uddevalla Hospital (Unknown); Skane University Hospital (Other); Lund University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTG1_081119
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Hepatitis C, Genotype 1
Keywords: Hepatitis C virus; Real-time PCR; Treatment
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Active Comparator): Treatment with Pegasys 180 µg/week and ribavirin 1000/1200 mg per day. Treatment is given for 24, 48 or 72 weeks depending on the time point (week 4, 12 or 24) when HCV RNA becomes undetectable by the Cobas Taqman assay. If HCV RNA has not declined 2 logs by week 12 or is detectable at week 24, treatment is stopped.
  Interventions: Drug: Peg-interferon-alfa2a (Pegasys); Drug: Ribavirin (Copegus)
- Tailored treatment (Experimental): Treatment with Pegasys 180 µg/week and ribavirin 1000/1200 mg per day. Treatment duration is flexible, 24-72 weeks, depending on the time point when the HCV RNA level is calculated to be 1 copy/mL. If the decline between day 14 and 28 is poor, treatment is stopped after 5 weeks.
  Interventions: Drug: Peg-interferon-alfa2a (Pegasys); Drug: Ribavirin (Copegus)

INTERVENTIONS:
Drug: Peg-interferon-alfa2a (Pegasys) — Peg-interferon-alfa2a 180 µg per week
  Other Names: Pegasys
Drug: Ribavirin (Copegus) — Ribavirin 1000 or 1200 mg per day depending on if body weight is below or above 75 kg

SUMMARY:
The purpose of the study is to investigate if the duration of treatment of hepatitis C with pegylated interferon and ribavirin can be individualized on the basis of how fast the hepatitis C virus concentration in the blood decreases, and if this is more cost-efficient than standard treatment.

DETAILED DESCRIPTION:
The current standard regimen for patients with chronic hepatitis C virus (HCV) infection, i.e., 48 weeks of pegylated interferon and ribavirin, needs to be further improved because of high costs and side-effects; in addition, the treatment is curative in only 50% of patients with genotype 1 of HCV. According to the current guidelines treatment with pegylated interferon and ribavirin is given for 24, 48 or 72 weeks depending on the time point when HCV-RNA becomes undetectable (week 4, 12 or 24). Patients with a very poor response may also be identified by applying a stopping rule at week 12 and 24. Still, most patients are treated for 48 weeks and a substantial number of those relapse after discontinuation.

In this study, standard treatment is compared with "tailored treatment", when the treatment duration is based on the time point when HCV RNA level is calculated to be 1 copy/mL, according measurements of HCV RNA on day 14, 21, 28 and 49. This arm also includes an earlier stopping rule: If the HCV RNA does not decline significantly between day 14 and 28, treatment is stopped after 5 weeks.

The advantage of tailored treatment is hypothesised to be that unnecessary side-effects and costs are avoided by an earlier identification of non-response and a treatment duration that is optimised for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Anti-HCV positive for > 6 months
* Genotype 1
* Clinical indication for treatment, preferably a liver biopsy showing significant inflammation and/or fibrosis
* Negative pregnancy test (for fertile women)

Exclusion Criteria:

* Pregnancy or breast-feeding
* Antiviral or immune modulating treatment the last 6 months
* Hepatitis B or HIV infection (HBsAg, anti-HIV)
* Other significant chronic liver disease
* History of bleeding esophageal varices or other signs of decompensation
* Neutrophiles < 1.0 x 109/L or platelets < 50 x 109/L. S-creatinine > 2 x ULN
* History of severe psychiatric disorder
* Autoimmune disease, severe heart disease, previous organ or stem cell transplantation, malignancy, thyroid disease, severe retinopathy
* Drug abuse, current or during the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-11; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Medication dose per cured patient | 26 weeks after end of treatment

SECONDARY OUTCOMES:
Sustained virological response and relapse rate | 26 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Lindh, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Background] Lindh M, Alestig E, Arnholm B, Eilard A, Hellstrand K, Lagging M, Wahlberg T, Wejstal R, Westin J, Norkrans G. Response prediction and treatment tailoring for chronic hepatitis C virus genotype 1 infection. J Clin Microbiol. 2007 Aug;45(8):2439-45. doi: 10.1128/JCM.00577-07. Epub 2007 Jun 20. PMID 17581934